CLINICAL TRIAL: NCT06452641
Title: Comparative Effects of Jones Technique and Cross Friction Massage on Pain, Range of Motion and Functional Disability in Patients With Cervicogenic Headache.
Brief Title: Effects of Jones Technique and Cross Friction Massage on Cervicogenic Headache.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/ RCR & AHS/23/01108
Record Dates: First submitted 2024-06-06; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Cervicogenic Headache
Keywords: Strain counter strain,; Cervicogenic Headache; neck pain; cross friction massage,
MeSH Terms: conditions — Post-Traumatic Headache; Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jones technique (Experimental): Strain counter strain (Jones technique) will be applied to this group
  Interventions: Other: Jones technique
- Cross-friction massage (Active Comparator): Cross-friction massage will be applied to this group.
  Interventions: Other: Cross-friction massage

INTERVENTIONS:
Other: Jones technique — Strain counter strain technique also known as Jones technique will be performed with the patient lay supine on the treatment table, taking them to a position-of-comfort by extending, side-bending, and rotating the head away (ESARA) from the TP until the TP pain has reduced. Continues to monitor, maintaining the patient's position for 90 seconds. After 90 seconds has elapsed, the patient's head should be slowly and passively returned to a neutral position with 3 sessions/week for 6 weeks. In essence, the TP should be relieved by placing the patient in a position of comfort, holding this position for 90 seconds, and slowly returning the patient to a neutral position.
  Arms: Jones technique
Other: Cross-friction massage — Group B will get cross friction massage for 15-20 mins. Participants will be treated 3 times per week for 6 weeks. Pre and Post-treatment readings will be taken in 1st session and 6th week respectively.
  Arms: Cross-friction massage

SUMMARY:
Cervicogenic headache is a very incessant issue that is often faced by the general population. Cervicogenic headache is a significant issue in patients with upper cervical dysfunction. However, its physical therapy management is a subject of debate. As the Comparative effects of Jones technique and cross-friction massage have never been investigated in patients with cervicogenic headache and neck pain, this study aims to investigate the effects of these treatments on two study groups (Group A&B) respectively.

DETAILED DESCRIPTION:
This study will be a randomized clinical trial and will be conducted in Al-Khidmat Foundation Sahiwal. The study will be completed within the time duration of six months. A nonprobability convenience sampling technique will be used to collect the data. The sample size of 30 patients will be taken in this study, aged 20-to 50 years, will be allocated to two groups, Group A (Jones technique) and Group B (cross friction massage). Strain counter strain technique also known as the Jones technique will be performed with the patient laid supine on the treatment table, taking them to a position of comfort by extending, side-bending, and rotating the head away (ESARA) from the TP until the TP pain has reduced. Continues to monitor, maintaining the patient's position for 90 seconds. After 90 seconds have elapsed, the patient's head should be slowly and passively returned to a neutral position with 3 sessions/week for 6 weeks.

Group B will get cross friction massage for 15-20 minutes. Participants will be treated 3 times per week for 6 weeks. Pre and Post-treatment readings will be taken in 1st session and 6th week respectively. Assessment will be done via a 6-item Headache Impact scale and neck disability index. The Neck Disability Index will be used to examine neck pain intensity and cervicogenic headache symptoms. The 6-item Headache Impact Test scale will be used to examine headache severity and its adverse effects on social life and functions. A goniometer will be used to assess the rotation range of motion.

ELIGIBILITY:
Inclusion Criteria:

* Headache with neck stiffness and/or pain.
* Headache for the past 3 months at least once per week
* Aged 20-40 years
* Chronic neck pain for more than 3 months
* Baseline NDI score of at least 20% (10 points).
* Forward head posture

Exclusion Criteria

* Headache with neck stiffness and/or pain.
* Headache for the past 3 months at least once per week
* Aged 20-40 years
* Chronic neck pain for more than 3 months
* Baseline NDI score of at least 20% (10 points).
* Forward head posture

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Pain: Visual Analogue Scale(VAS) | 4th week
  A Visual Analogue Scale (VAS) is one of the pain rating scales used for the first time in 1921 by Hayes and Patterson. It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms. From the patient's perspective, this spectrum appears continuous; their pain does not take discrete jumps, as a categorization of none, mild, moderate and severe would suggest. It was to capture this idea of an underlying continuum that the VAS was devised.
Function: Headache Impact Test - HIT-6 | 4th week
  The HIT-6 consists of six items: pain, social functioning, role functioning, vitality, cognitive functioning, and psychological distress. The patient answers each of the six related questions using one of the following five responses: "never", "rarely", "sometimes", "very often", or "always".
Active cervical range of motion | 4th week
  To measure the cervical range of motion, the universal goniometer will use
Disability: Neck Disability Index NDI | 4th week
  The Neck Disability Index (NDI) is a 10-item questionnaire that measures a patient's self-reported neck pain related disability. A higher NDI score means the greater a patient's perceived disability due to neck pain. The minimally clinically important change by patients has been found to be 5 or 10%.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Hajra, Principal Investigator — Riphah International University
Locations (1):
- Al-Khidmat foundation Sahiwal., Sahiwal, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ylinen J, Nikander R, Nykanen M, Kautiainen H, Hakkinen A. Effect of neck exercises on cervicogenic headache: a randomized controlled trial. J Rehabil Med. 2010 Apr;42(4):344-9. doi: 10.2340/16501977-0527. PMID 20461336
- [Background] Mohamed AA, Shendy WS, Semary M, Mourad HS, Battecha KH, Soliman ES, Sayed SHE, Mohamed GI. Combined use of cervical headache snag and cervical snag half rotation techniques in the treatment of cervicogenic headache. J Phys Ther Sci. 2019 Apr;31(4):376-381. doi: 10.1589/jpts.31.376. Epub 2019 Apr 1. PMID 31037013
- [Background] Yang DJ, Kang DH. Comparison of muscular fatigue and tone of neck according to craniocervical flexion exercise and suboccipital relaxation in cervicogenic headache patients. J Phys Ther Sci. 2017 May;29(5):869-873. doi: 10.1589/jpts.29.869. Epub 2017 May 16. PMID 28603362
- [Background] Watson DH, Trott PH. Cervical headache: an investigation of natural head posture and upper cervical flexor muscle performance. Cephalalgia. 1993 Aug;13(4):272-84; discussion 232. doi: 10.1046/j.1468-2982.1993.1304272.x. PMID 8374943
- [Background] Putra IPM, Nugraha MHS, Tianing NWJPTJoI. Combined Deep Transverse Friction and Muscle Energy Technique on Mechanical Neck Pain: Article Review. 2020;1(1):17-22.
- [Background] Khan ZK, Ahmed SI, Baig AAM, Farooqui WA. Effect of post-isometric relaxation versus myofascial release therapy on pain, functional disability, rom and qol in the management of non-specific neck pain: a randomized controlled trial. BMC Musculoskelet Disord. 2022 Jun 13;23(1):567. doi: 10.1186/s12891-022-05516-1. PMID 35698187
- [Background] Yasin M, Gondal MJI, Qamar MM, Basharat A, Rasul A, Ahmed WJMJoDDPU. Effects of deep friction massage and static stretching in non-specific neck pain. 2019;12(4):331-4.
- [Background] Kong YS, Kim YM, Shim JM. The effect of modified cervical exercise on smartphone users with forward head posture. J Phys Ther Sci. 2017 Feb;29(2):328-331. doi: 10.1589/jpts.29.328. Epub 2017 Feb 24. PMID 28265167